CLINICAL TRIAL: NCT05603312
Title: A Randomized, Double-Blind, Sham-Controlled Study to Evaluate the Safety and Tolerability of Glutamic Acid Decarboxylase Gene Transfer to the Subthalamic Nuclei in Participants With Parkinson's Disease
Brief Title: A Double-blind Study to Evaluate the Safety of Glutamic Acid Decarboxylase Gene Transfer in Parkinson's Participants
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MeiraGTx, LLC (Industry)
Responsible Party: Sponsor
Organization: MeiraGTx UK II Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MGT-GAD-025
Record Dates: First submitted 2022-10-12; First posted 2022-11-02 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Participants are enrolled in one of three groups in parallel for the duration of the study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (3):
- AAV-GAD Low Dose (Experimental): Eligible participants received bilateral infusion of AAV-GAD low dose into the STN
  Interventions: Genetic: AAV-GAD Low Dose
- AAV-GAD High Dose (Experimental): Eligible participants received bilateral infusion of AAV-GAD high dose into the STN
  Interventions: Genetic: AAV-GAD High Dose
- Sham Surgery (Sham Comparator): Eligible participants underwent a sham surgical procedure
  Interventions: Procedure: Sham Surgery

INTERVENTIONS:
Genetic: AAV-GAD Low Dose — Bilateral infusion of AAV-GAD low dose
  Arms: AAV-GAD Low Dose
Genetic: AAV-GAD High Dose — Bilateral infusion of AAV-GAD high dose
  Arms: AAV-GAD High Dose
Procedure: Sham Surgery — Sham infusion
  Arms: Sham Surgery

SUMMARY:
The objective of this clinical trial was to evaluate the safety and tolerability of adeno-associated virus (AAV)-mediated delivery of glutamic acid decarboxylase (GAD) gene transfer into the subthalamic nuclei (STN) of participants with Parkinson's Disease.

DETAILED DESCRIPTION:
The planned length of participation in the study for each participant was approximately 7 months, including a screening period of up to 40 days, randomization, surgery, and a follow-up period of 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Parkinson's Disease
* Levodopa responsiveness for at least 12 months
* UPDRS Part 3 score of ≥25 points in the "off" state

Exclusion Criteria:

* History of brain surgery to treat Parkinson's Disease
* Any history of cerebral insult or central nervous system infection
* Atypical Parkinson's Disease
* Focal or lateralized neurologic deficits
* Evidence of significant medical or psychiatric disorders
* Cognitive impairment as defined by the Montreal Cognitive Assessment (MoCA) ≤ 20
* Beck Depression Inventory-II score of ≥ 20

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Yale University - Yale New Haven Hospital, New Haven, Connecticut
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Weill Cornell Medicine, New York, New York
  - Columbia University Irving Medical Center, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 6 medical centers in the United States (US). A total of 14 participants were enrolled in the study.
Groups:
- AAV-GAD Low Dose: Bilateral infusion of AAV-GAD Low Dose into the STN
- AAV-GAD High Dose: Bilateral infusion of AAV-GAD High Dose into the STN
Period: Overall Study
Arm/Group | AAV-GAD Low Dose | AAV-GAD High Dose | Sham Surgery
Started | 5 | 5 | 4
Completed | 5 | 5 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AAV-GAD Low Dose | AAV-GAD High Dose | Sham Surgery | Total
Number analyzed (Participants) | 5 | 5 | 4 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 2 | 5
  >=65 years | 4 | 3 | 2 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 3
  Male | 4 | 3 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 4 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 5 | 4 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 4 | 14

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events Related to the Treatment
Description: The primary outcome measure is the safety of treatment with AAV-GAD, assessed by the absence of IMP-related treatment-emergent adverse events.
Time Frame: Baseline to Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | AAV-GAD Low Dose | AAV-GAD High Dose | Sham Surgery
Number analyzed (Participants) | 5 | 5 | 4
Participants | 0 | 1 | 0

2. Primary Outcome: Incidence of Serious Adverse Events Related to the Treatment
Description: The primary outcome measure is the safety of treatment with AAV-GAD, assessed by the absence of IMP-related serious treatment-emergent adverse events.
Time Frame: Baseline to Week 26
Measure: Count of Participants; unit: Participants
Arm/Group | AAV-GAD Low Dose | AAV-GAD High Dose | Sham Surgery
Number analyzed (Participants) | 5 | 5 | 4
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From the signing of the Informed Consent Form to Week 26
Description: Safety was evaluated by vital signs, neurological and physical examinations, electrocardiograms, radiographic imaging, and clinical laboratory tests.
  Treatment-related AEs were reported in 1 participant. This participant (high-dose group) experienced mild confusion and a mild headache perioperatively. These events started on the day of surgery and resolved the same day and 11 days later, respectively. All other AEs and all SAEs were assessed by the Investigator as unrelated to the study drug.
Arm/Group | AAV-GAD Low Dose | AAV-GAD High Dose | Sham Surgery
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/5 | 1/4
Other Adverse Events (participants affected / at risk) | 5/5 | 5/5 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AAV-GAD Low Dose (N=5) | AAV-GAD High Dose (N=5) | Sham Surgery (N=4)
Catheter site haemorrhage (General disorders) | 1 | 0 | 0
Freezing phenomenon (Nervous system disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AAV-GAD Low Dose (N=5) | AAV-GAD High Dose (N=5) | Sham Surgery (N=4)
Palpitations (Cardiac disorders) | 0 | 1 | 0
Eye swelling (Eye disorders) | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Fatigue (General disorders) | 1 | 2 | 0
Gait disturbance (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 1
Confusion postoperative (Injury, poisoning and procedural complications) | 1 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Computerised tomogram abnormal (Investigations) | 1 | 1 | 0
Haematocrit decreased (Investigations) | 0 | 1 | 0
Red blood cells urine positive (Investigations) | 0 | 0 | 1
Reflex test abnormal (Investigations) | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 1 | 1
Facial spasm (Nervous system disorders) | 0 | 1 | 0
Head discomfort (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 3 | 0
Hyperreflexia (Nervous system disorders) | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
On and off phenomenon (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 1
Thrombophlebitis (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT05603312/Prot_SAP_000.pdf